CLINICAL TRIAL: NCT03422991
Title: Lyon and Rhône Alpes Auvergne Registry of Congestive Heart Failure
Brief Title: Cohort of Heart Failure Patients
Acronym: LOOP-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0250
Record Dates: First submitted 2018-01-12; First posted 2018-02-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Cohort
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases; Vascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Congestive Heart Failure patients Cohort (Other): Cluster of patients with congestive heart failure NYHA ≥2, with at least one cardiac decompensation, NT-proBNP (N-terminal pro-brain natriuretic peptide) > 500 ng/l. Will be followed during 18 months.
  Interventions: Other: Blood sampling and Quality of life questionnaire.

INTERVENTIONS:
Other: Blood sampling and Quality of life questionnaire. — Blood sampling and Quality of life questionnaire.

SUMMARY:
This is a prospective cohort study of patients with Heart Failure with an eighteen-month follow-up aimed to collect all demographic, clinical, biological and para-clinical data to study population characteristics, assess prognosis markers and occurrence of HF treatment side effects.

Congestive Heart failure is a frequent pathology and its prevalence increases with age. Its prognosis stays pejorative despite years of major therapeutical progress. In recent trials, all-cause mortality rates at 1-year reach up to 20% and 50% at 5 years.

Medical care of congestive heart failure is based on precise international recommendations. The association of Beta-Blockers, renin-angiotensin system blockers, mineralocorticoid receptor antagonists, represent the basis of the pharmacological treatment.

Cardiac resynchronization treatment and implantable cardioverter-defibrillator are additional efficient treatments that reduce events in appropriately selected patients.

Despite these improvements, the prognostic of congestive heart failure in registers is worse than those observed in randomized trials. This can be explained by differences in congestive heart failure patient populations and/or by a less rigorous medical care where treatments are not optimized.

The evaluation of medical care in congestive heart failure is today of utmost importance.

Integrating new pharmacological molecules, medical devices and the application of new recommendations have major interest for documentation and practical changes.

The main objective of this cohort will be to evaluate the evolution of the 12-month quality of life score of a HF patient and the characteristics and treatments associated with it.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congestive heart failure confirmed during

  * Hospitalization for cardiac decompensation
  * A medical follow-up for stable congestive heart failure with at least one cardiac decompensation event
* NT-proBNP > 500 ng/l in the month before Baseline (or BNP > 150 ng/l)
* NYHA ≥ 2
* Aged over 18
* Signature of the informed consent

Exclusion Criteria:

* Life expectancy shorter than a month
* Patients on long term assistance or with heart transplant
* Impossibility to give patients clear information
* Loss of autonomy, dementia, major dependence
* Patients without health coverage
* Patient with no legal protection
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Quality of life questionnaire : EuroQol (EQ-5D) at 12 months | 12 months
  Measurement of quality of life of patients with heart failure: patient will answer to this questionnaire (Mobility, Autonomy of the person, Current activities, Pain ,Anxiéty/Depression)
  ) at baseline and at 12th month visit. The evolution between these two scores will be analysed .

SECONDARY OUTCOMES:
Renal function : glomerular filtration rate | Baseline
  Assessing the renal function evolution of patients with heart failure the glomerular filtration rate will be calculated according to CKD-EPI (Chronic Kidney Disease - Epidemiology Collaboration) formula.
Renal function : glomerular filtration rate | 2 months
  Assessing the renal function evolution of patients with heart failure the glomerular filtration rate will be calculated according to CKD-EPI (Chronic Kidney Disease - Epidemiology Collaboration) formula.
NT-proBNP | 18 months
  Measure of NT-proBNP will be done at 18th month in order to correlate the effect of low blood pression and renal function decreasing on NT-proBNP variability
number of death (all-cause) | 18 months
number of all cardiovascular cause death | 18 months
number all unscheduled hospitalization for heart failure | 18 months
number of stroke | 18 months
nonfatal myocardial infarction | 18 months
cardiac assistance or heart transplantation | 18 months
symptomatic hypotension | 18 months
number of dialysis | 18 months
number ventricular arrhythmias | 18 months
  (ventricular tachycardia and ventricular fibrillation)
Heart failure stage will be assessed thanks to the New York Heart Association (NYHA) classification | Baseline, 6, 12 and 18 months
Cardiac function | Baseline and 12 months
  Cardiac function will be evaluated on Echography Trans Thoracic at baseline and at the 12 months visit.
  * Left Ventricular Ejection Fraction
  * levitation pressure filling (yes/No)
  * Right ventricular dysfunction (yes/no)
  * pulmonary artery systolic pressure (mmHg)
  * right atrial pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Louis Pradel, Centre d'Investigation Clinique, Lyon, France

IPD SHARING:
Plan to Share IPD: No